CLINICAL TRIAL: NCT06733623
Title: Does the Presence and Type of Curves Influence the Choice of Asymmetric Postures Adopted in Daily Life by Patients with Juvenile and Adolescent Idiopathic Scoliosis?
Brief Title: Impact of Spinal Curves on Asymmetric Posture in Idiopathic Scoliosis
Acronym: ISAPIS
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Scientifico Italiano Colonna Vertebrale (Other)
Responsible Party: Sponsor
Other Study IDs: 5461_20.11.2024_P_bis
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS); Juvenile Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Scoliosis patients: Patients aged between 6 and 18 years old with a diagnosis of idiopathic scoliosis are asked to answer a questionnaire investigating the preferred postures adopted daily
- Control group: Subjects aged between 6 and 18 years old without a diagnosis of idiopathic scoliosis are asked to answer a questionnaire investigating the preferred postures adopted daily

SUMMARY:
Asymmetric postures are often observed in patients with adolescent idiopathic scoliosis (AIS) and are partially associated with instability in sitting and standing positions, as well as with imbalances in gait kinematic parameters in cases of moderate or severe scoliosis.

Based on the currently available data, no correlation has been identified between habitual postures in daily life and the presence of scoliosis. However, the asymmetry of preferred postures in relation to the morphological characteristics of the curves, and how this might contribute to the progression of the clinical condition due to prolonged uneven load distribution, has not yet been analyzed.

Understanding any preferential direction in postures habitually adopted by patients with idiopathic scoliosis could provide valuable insights for the conservative management of the condition.

The aim of this study is to analyze the influence of the morphological characteristics of scoliotic curves (type and laterality) in patients with juvenile and adolescent idiopathic scoliosis on the choice of preferentially maintained asymmetric postures in daily life, using a descriptive questionnaire completed by family members and caregivers, compared to a group of non-scoliotic subjects.

Evaluate the effect of curve magnitude, age, sex, and Risser grade on the choice of usual asymmetric postures.

Estimate the impact of prolonged maintenance of habitual asymmetric postures on the clinical progression in patients with juvenile and adolescent idiopathic scoliosis

ELIGIBILITY:
Scoliosis group:

Inclusion Criteria:

* Diagnosis of juvenile or adolescent idiopathic scoliosis;
* Age between 6 and 18 years;
* Full spine X-ray in a standing position with anteroposterior projection performed within the year prior to completing the questionnaire.

Exclusion Criteria:

* Diagnosis of secondary scoliosis
* Patients with neuromotor control disorders

Control group:

Inclusion criteria:

* Age between 6 and 18 years;
* No diagnosis of sciolisis
* Full spine X-ray in a standing position with anteroposterior projection performed within the year prior to completing the questionnaire.

Exclusion Criteria:

- Patients with neuromotor control disorders

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The participants of the study are patients of a tertiary referral outpatient clinic specializing in the conservative treatment of spinal deformity
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Everyday posture questionnaire | At enrollment
  The types of postures most frequently maintained in daily life by patients with idiopathic scoliosis will be compared with a group of age-matched individuals without scoliosis, and any statistically significant differences will be analyzed using the chi-square test

CONTACTS AND LOCATIONS:
Locations (1):
- ISICO, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be uploaded on a public repository (Zenodo)